CLINICAL TRIAL: NCT06315322
Title: A MULTICENTER, OPEN-LABEL, SINGLE-ARM STUDY TO EVALUATE LONG-TERM SAFETY AND TOLERABILITY OF BRIVARACETAM IN STUDY PARTICIPANTS WITH CHILDHOOD ABSENCE EPILEPSY OR JUVENILE ABSENCE EPILEPSY
Brief Title: A Study to Test the Long-term Safety and Tolerability of Brivaracetam in Study Participants With Childhood Absence Epilepsy or Juvenile Absence Epilepsy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP0224; 2023-508095-11-00 (Registry Identifier: EU Trial Number); U1111-1303-1174 (Other: Universal Trial Number)
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Childhood Absence Epilepsy; Juvenile Absence Epilepsy
Keywords: Childhood Absence Epilepsy; Juvenile Absence Epilepsy; Phase 3; Brivaracetam
MeSH Terms: conditions — Epilepsy, Absence | interventions — brivaracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Brivaracetam arm (Experimental): Subjects in this arm will receive various brivaracetam doses as oral solution or film-coated tablet twice per day.
  Interventions: Drug: Brivaracetam Film-coated tablet; Drug: Brivaracetam oral solution

INTERVENTIONS:
Drug: Brivaracetam Film-coated tablet — Drug: Brivaracetam Film-coated tablet Pharmaceutical form: Film-coated tablet Route of administration: Oral use Brivaracetam film-coated tablet [10, 25 or 50 mg] will be administered twice per day in equal doses.
Drug: Brivaracetam oral solution — Pharmaceutical form: Oral solution Route of administration: Oral use Brivaracetam oral solution [10 mg/mL]) will be administered twice per day in equal doses.

SUMMARY:
The purpose of the study is to investigate the long-term safety and tolerability of brivaracetam in study participants with childhood absence epilepsy or juvenile absence epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Participants who previously participated in EP0132 (NCT05109234) and/or N01269 (NCT04666610) and qualify for entry into EP0224 as per the EP0132 or N01269 protocol with a confirmed diagnosis of childhood absence epilepsy (CAE) or juvenile absence epilepsy (JAE)
* Participants for whom a reasonable benefit from long-term administration of Brivaracetam (BRV) is expected in the opinion of the Investigator
* Male and female A male participant must agree to use contraception during the treatment period and for at least 2 days after the final dose of investigational medicinal product (IMP) and refrain from donating sperm during this period.

A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

◦ Not a woman of childbearing potential (WOCBP) OR A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 2 days after the final dose of IMP.

- Capable of and provides informed consent/assent, and the participant's parent/legal representative/caregiver provides signed informed consent for minor participants, which includes compliance with the requirements and restrictions listed in the Informed Consent form (ICF)/Assent form and in this protocol

Exclusion Criteria:

* Participant has a history or presence of paroxysmal nonepileptic seizures
* Participant has severe medical, neurological, or psychiatric disorders or laboratory values which could, at the discretion of the Investigator, affect safe participation in the study or would preclude appropriate study participation
* Participant has hepatic impairment (Child Pugh Score A, B, or C) based on the Investigator's assessment
* Participant has active suicidal ideation prior to study entry as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) (for participants 6 years of age or older) or clinical judgment (for participants younger than 6 years of age). The participant should be referred immediately to a Mental Healthcare Professional
* Participant has any medical or psychiatric condition that, in the opinion of the Investigator, could jeopardize or would compromise the participant's ability to participate in this study
* Participant has known fructose intolerance or a known hypersensitivity to any components of BRV or excipients or a drug with similar chemical structure
* Concomitant use of carbamazepine, felbamate, gabapentin, oxcarbazepine, phenobarbital, phenytoin, tiagabine, or vigabatrin
* Participant is receiving any investigational drugs or using any experimental devices in addition to BRV
* Participant meets a mandatory withdrawal criterion for N01269 or EP0132 or is experiencing an ongoing Serious adverse event (SAE)
* Participant has poor compliance with the visit schedule or IMP intake in the preceding study in the opinion of the Investigator

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2030-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) during the study | From Entry Visit up to the Safety Visit (up to 3 years)
  An adverse event (AE) is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory finding) in study participants, users, or other persons, whether or not related to the investigational medicinal product (IMP).
Incidence of treatment-emergent adverse events (TEAEs) leading to discontinuation of investigational medicinal product (IMP) during the study | From Entry Visit up to the Safety Visit (up to 3 years)
  An adverse event (AE) is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory finding) in study participants, users, or other persons, whether or not related to the investigational medicinal product (IMP).

SECONDARY OUTCOMES:
Incidence of serious adverse events (SAEs) during the study | From Entry Visit up to the Safety Visit (up to 3 years)
  A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires in patient hospitalization or prolongation of existing hospitalization
  * Is a congenital anomaly or birth defect
  * Results in permanent or significant disability/incapacity
  * Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above
Incidence of IMP related TEAEs during the study | From Entry Visit up to the Safety Visit (up to 3 years)
  An adverse event (AE) is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory finding) in study participants, users, or other persons, whether or not related to the investigational medicinal product (IMP).

CONTACTS AND LOCATIONS:
Locations (23):
- United States (5):
  - Ep0224 50140, Birmingham, Alabama
  - Ep0224 50639, Orange, California
  - Ep0224 50268, Miami, Florida
  - Ep0224 50638, New Brunswick, New Jersey
  - Ep0224 50640, Winston-Salem, North Carolina
- Georgia (4):
  - Ep0224 20321, Tbilisi
  - Ep0224 20322, Tbilisi
  - Ep0224 20323, Tbilisi
  - Ep0224 20324, Tbilisi
- Italy (6):
  - Ep0224 40144, Abbiategrasso
  - Ep0224 40765, Messina
  - Ep0224 40764, Pavia
  - Ep0224 40629, Roma
  - Ep0224 40766, Roma
  - Ep0224 40763, Verona
- Romania (4):
  - Ep0224 40767, Bucharest
  - Ep0224 40769, Bucharest
  - Ep0224 40768, Iași
  - Ep0224 40770, Timișoara
- Slovakia (2):
  - Ep0224 40771, Bardejov
  - Ep0224 40772, Dubnica nad Váhom
- Ep0224 40453, Terrassa, Spain
- Ep0224 20328, Uzhhorod, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://vivli.org/